CLINICAL TRIAL: NCT04486092
Title: Mood Stabilizer-induced Metabolic Abnormalities in Bipolar Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-ER-104-031
Record Dates: First submitted 2015-10-11; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-01

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Valproic Acid

ARMS (1):
- Valproic Acid (Experimental)
  Interventions: Drug: Valproic Acid

INTERVENTIONS:
Drug: Valproic Acid

SUMMARY:
The potential effects of microbiota in bipolar disorder (BD) with microbiota-related dysfunction have not yet been explored clinically, and the integration of microbiota and pharmacometabolomic approaches can provide us the identification of the significant effects of mood stabilizers on metabolic homeostasis, treatment response, and cognitive performance. Therefore, we propose to develop the integration of the microbiota and pharmacometabolomics knowledge base about the mood stabilizer-induced metabolic abnormalities in BD patients.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar disorder outpatients (aged 18-65 years) who meet the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) diagnostic criteria and start to receive valproate (VPA) will be enrolled consecutively by trained psychiatrists.

Exclusion Criteria:

* Exclude are patients who had DSM-V diagnosis for substance abuse within the past three months
* Had treated with antibiotics and/or functional foods (probiotics and/or prebiotics) for at least one month before entering study
* Presence of stomach/gut problems such as chronic diarrhea, constipation, gas, heartburn, bloating, etc.
* Had an organic mental disorder, mental retardation, dementia, or other diagnosed neurological illness
* Had a surgical condition or a major physical illness
* Were pregnant or breast-feeding
* Had any concomitant DSM-V Axis I diagnoses together with somatic or neurologic illnesses interfering psychiatric evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-02; Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota composition | 12 weeks

SECONDARY OUTCOMES:
Metabolic syndrome | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University (NCKU) Hospital, Tainan, Taiwan